CLINICAL TRIAL: NCT05827731
Title: Study on the Factors Influencing the Delivery Mode of Pregnant Women Induced by Cervical Double Balloon Combined With Oxytocin
Brief Title: Cervical Double Balloon Combined With Oxytocin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changsha Hospital for Maternal and Child Health Care (Other)
Responsible Party: Principal Investigator, Qiu-Hong Xiang, Principal investigator, Changsha Hospital for Maternal and Child Health Care
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ChangshaHMC 331
Record Dates: First submitted 2023-04-05; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy Outcomes; Oxytocin; Labor Induction; Mode of Delivery
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural delivery group (No Intervention): The patients in this group were treated with natural delivery
- Cesarean section group (Experimental): The patients in this group were delivered by cesarean section
  Interventions: Behavioral: cesarean section

INTERVENTIONS:
Behavioral: cesarean section — According to the different outcomes of pregnancy, the patients were divided into natural delivery group and cesarean section group
  Arms: Cesarean section group

SUMMARY:
1 Materials and methods 1.1 Subjects From September 2021 to August 2022, the patients who received induction of labor by cervical double balloon combined with oxytocin in a Grade III A Maternal and Child Health Hospital in Changsha were included in the study. A double balloon and oxytocin induced labor at a tertiary maternal and child health centre in Changsha. Inclusion criteria: 1 age ≥18 years; 2 Singleton; 3 no vaginal infection, fetal membranes intact; 4 according with the indication of induced labor [5] ; These included delayed pregnancy, hypertensive disorder complicating pregnancy, diabetes mellitus, cervical Bishop score < 6, and negative oxytocin provocation test (Oct) . The exclusion criteria were: 1 abnormal head and pelvis, unable to be delivered vaginally; 2 twins; 3 maternal contraindication of vaginal delivery; 4 severe placental dysfunction, unable to tolerate vaginal delivery; 5 there were contraindications for the use of cervical balloon.

1.2 Methods 1.2.1 Operation Method First of all, pregnant women to introduce the procedure of placing the balloon, ease their fear, tension. Assist the patient to take the stone position, sterilize vulva 3 times, spread aseptic towel, expose cervix with vaginal speculum, sterilize vagina and cervix 3 times with iodine cotton ball, after sterilizing the cervical tube 3 times with iodine-complexed cotton swab, insert the disposable dilatation balloon (Henan Bonding Industry Co., Ltd., Yusheng Medical Supervision Machine No. 20180029, model: Type II 18F) into the cervical tube, until the two sacs into the cervical canal and ensure that the double sacs are through the cervical mouth, sub-turn to the cervical inside and outside sacs slowly injected saline 80 ml each. The end of the balloon catheter was fixed to the inner thigh of the pregnant woman with 3m adhesive tape, without restricting the physical activity of the pregnant woman. The operation process is smooth, the pregnant woman has no discomfort, before and after the operation monitoring fetal heart is normal, instructs the pregnant woman to test the fetal movement, closely observes the pregnant woman labor sign and the fetal intrauterine situation. The balloon is usually inserted between 16:00 and 18:00. The balloon is taken out at 8:00 am the next day, oxytocin (Ringe 500ml + oxytocin 2.5 U) was given intravenously to the patients who were not in Labor 1 hour after rupture of membranes. According to the frequency of uterine contractions, if there is no uterine contractions, increase the rate of dripping 8 drops/min, maximum dose not more than 40 drops, until regular uterine contractions, after every half-hour assessment.

1.2.2 Observation indicators Using the hospital electronic medical record information system to search and review the medical records of these women, the age, number of pregnancies, number of parturients, weight gain during pregnancy, height, weight, pre-and post-pregnancy body mass index (BMI) , indication of induced labor, pregnancy complications, gestational age at the time of balloon induced labor, neonatal weight, cervical Bishop score before and after balloon dilatation, occurrence of acute Chorioamnionitis, fetal distress, NST typing, mode of delivery, etc. . The clinical data of the patients who were induced by cervical double balloon combined with oxytocin were analyzed, and the related factors of pregnancy outcome were also discussed.

1.3 Statistical credits SPSS 25.0 was used to analyze the data. The mean ± standard deviation was used for statistical description and t-test was used for statistical analysis. The frequency was used for statistical description and chi-square test was used for statistical analysis. Binary logistic regression analysis was used to determine the influencing factors of different pregnancy modes, and the difference was statistically significant with P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* Singleton
* no vaginal infection, fetal membranes intact
* according with the indication of induced labor [5] ; These included delayed pregnancy, hypertensive disorder complicating pregnancy, diabetes mellitus, cervical Bishop score < 6, and negative oxytocin provocation test (Oct)

Exclusion Criteria:

* abnormal head and pelvis, unable to be delivered vaginally
* twins
* maternal contraindication of vaginal delivery
* severe placental dysfunction, unable to tolerate vaginal delivery
* there were contraindications for the use of cervical balloon.

Ages: 25 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Acute Chorioamnionitis | Immediately after the surgery
  acute Chorioamnionitis (or = 0.006,95% cl = 0.001-0.030, p < 0.001)
Fetal distress | Immediately after the surgery
  fetal distress (or = 0.102,95% CL = 0.022-0.473, P = 0.004)
NST typing | Immediately after the surgery
  NST typing (or = 20.057,95% CL = 4.145-97.039, p < 0.001)

CONTACTS AND LOCATIONS:
Locations (1):
- Changsha Hospital for Maternal & Child Health Care Affiliated to Hunan Normal University, Changsha, Hunan, China